CLINICAL TRIAL: NCT00091039
Title: A Pilot Trial of a CEA/TRICOM-Based Vaccine in Combination With Combined Chemotherapy/Radiotherapy in Patients With Unresectable Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Vaccine Therapy, Chemotherapy, and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed With Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000383146; NCI-04-C-0252; NCI-6439; NCT00088725 (obsolete NCT alias)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: recombinant fowlpox GM-CSF vaccine adjuvant
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine
Biological: recombinant vaccinia-CEA(6D)-TRICOM vaccine
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high energy x-rays to damage tumor cells. Combining vaccine therapy with chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This clinical trial is studying how well giving vaccine therapy together with paclitaxel, carboplatin, and radiation therapy works in treating patients with stage III non-small cell lung cancer that cannot be removed with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of standard paclitaxel, carboplatin, and radiotherapy in combination with vaccinia-CEA-TRICOM vaccine, fowlpox-CEA-TRICOM vaccine, and recombinant fowlpox GM-CSF vaccine in patients with unresectable stage III non-small cell lung cancer.

Secondary

* Determine clinical response in patients treated with this regimen.
* Determine time to disease progression and overall median survival of patients treated with this regimen.
* Determine immunologic response in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Vaccine: Patients receive vaccinia-CEA-TRICOM vaccine subcutaneously (SC) on day 0 and fowlpox-CEA-TRICOM (rF-CEA-TRICOM) vaccine SC on days 14, 29, 43, 57, 70, 91, and 112. Patients also receive recombinant fowlpox GM-CSF (rF-GM-CSF) vaccine SC with each vaccination. Patients with stable or responding disease after day 112 continue to receive rF-CEA-TRICOM and rF-GM-CSF SC every 3 weeks in the absence of disease progression or unacceptable toxicity.
* Radiotherapy: Patients undergo radiotherapy on days 21-25, 28-32, 35-39, 42-46, 49-53, 56-60, and 63-67.
* Chemotherapy: Concurrently with radiotherapy, patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 21, 28, 35, 42, 49, 56, and 63. Patients also receive paclitaxel and carboplatin on days 91 and 112 (after completion of radiotherapy).

Patients are followed annually for up to 15 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 4-6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage III (locally advanced) disease
* Unresectable disease
* Carcinoembryonic antigen (CEA)-positive (staining ≥ 20% of cells) tumor by immunohistochemistry
* HLA-A2-positive
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Absolute lymphocyte count ≥ 600/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin < 1.5 mg/dL
* AST ≤ 2 times upper limit of normal
* Hepatitis B and C negative

Renal

* Creatinine normal OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No unstable or newly diagnosed angina pectoris
* No myocardial infarction within the past 6 months
* No New York Heart Association class II-IV congestive heart failure

Immunologic

* HIV negative
* No altered immune function
* No active or history of eczema
* No atopic dermatitis
* No autoimmune disease, including any of the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus
  * Sjögren's syndrome
  * Scleroderma
  * Myasthenia gravis
  * Goodpasture's syndrome
  * Addison's disease
  * Hashimoto's thyroiditis
  * Active Graves' disease
  * Multiple sclerosis
* No known history of allergy or serious reaction to prior vaccination with vaccina
* No known allergy to eggs
* No active or history of extensive psoriasis, severe acneiform rash, impetigo, varicella zoster, burns, or other traumatic or pruritic skin condition

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study participation
* No history of seizures or encephalitis
* Able to avoid close household contact with the following individuals for at least 3 weeks after vaccinia vaccination:

  * Children under 3 years of age
  * Pregnant or nursing women
  * Individuals with a history of or active eczema or other eczematoid skin disorders
  * Individuals with other acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, impetigo, burns, varicella zoster, severe acne, or other open rashes or wounds)
  * Immunodeficient or immunosuppressed individuals, including HIV-positive persons, by disease or therapy
* No other active malignancy within the past 2 years
* No other concurrent serious illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 years since prior immunotherapy with related vaccinia and fowlpox vaccines
* At least 3 years since prior antigen-specific peptides
* No other concurrent immunotherapy

Chemotherapy

* No prior paclitaxel or carboplatin for lung cancer
* At least 3 years since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent steroids, except for any of the following:

  * Topical steroids
  * Inhaled steroids for mild or moderate asthma
  * Dexamethasone as premedication for paclitaxel OR for short-term doses (48-72 hours in duration) to control refractory nausea that is not responding to other antiemetics
  * Systemic corticosteroids for ≥ grade 3 radiation pneumonitis
* No steroid eye-drops for at least 3 weeks after vaccinia vaccination
* No concurrent hormonal therapy
* No concurrent systemic glucocorticoids

Radiotherapy

* No prior radiotherapy to the lung fields
* No prior thoracic radiotherapy for lung cancer
* No other concurrent radiotherapy

Surgery

* Surgical scars must be healed
* No prior splenectomy
* No concurrent major surgical procedure

Other

* Recovered from all prior therapy
* No other concurrent anticancer agent or therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Arlen, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States